CLINICAL TRIAL: NCT03853863
Title: Walking With Minimalist Shoes to Promote Intrinsic Foot Muscle Growth and Foot Arch Integrity in Preschool Children: A Randomized Controlled Trial
Brief Title: Minimalist Shoes Walking for Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: Chinese University of Hong Kong (Other); Harvard Medical School (HMS and HSDM) (Other)
Responsible Party: Principal Investigator, Dr Roy Tsz-hei CHEUNG, Associate Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HMRF_RC
Record Dates: First submitted 2019-02-20; First posted 2019-02-26 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2019-08

CONDITIONS: Muscle Strength; Ultrasonography; Child, Preschool
Keywords: foot muscle strength; foot muscle size; minimal footwear; preschool child; ultrasonography

STUDY DESIGN:
Intervention Model Description: the single-blinded randomized control trial
Who Masked: Investigator
Masking Description: Assessment will be conducted by independent researchers who are not involved in subject allocation.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- minimalist shoes walking group (MSW) (Experimental): Subjects in the MSW group will be given a pair of minimalist shoes for all in-school activities (i.e., in-school walking training with minimalist shoes).
  Interventions: Behavioral: in-school walking training with minimalist shoes
- traditional shoes walking group (TSW) (Active Comparator): Subjects in the TSW group will be given a pair of protective shoes with arch support while following the same wearing pattern as the MSW group (i.e., in-school walking training with protective shoes).
  Interventions: Behavioral: in-school walking training with protective shoes

INTERVENTIONS:
Behavioral: in-school walking training with minimalist shoes — Participants in the MSW group will be given a pair of minimalist shoes for all in-school activities (i.e., 5 days/week and 7 hours/day) for 12 weeks. Similar to previous minimalist footwear studies, the intervention duration will be gradually increased over the 12-week training. In brief, subjects will wear the minimalist shoes for 1 out of 5 school days at the first week; 2 days at the second week, and so on until fully use of the minimalist shoes at the fifth week.
  Arms: minimalist shoes walking group (MSW)
Behavioral: in-school walking training with protective shoes — Participants in the TSW group will be given a pair of given a pair of protective shoes with arch support for all in-school activities (i.e., 5 days/week and 7 hours/day) for 12 weeks,while follow the same wearing pattern as the MSW group.
  Arms: traditional shoes walking group (TSW)

SUMMARY:
This is a single-blind randomized control study that will investigate the effects of a 12-week in-school walking training with minimalist shoes for local preschool children on intrinsic foot muscle size, muscle strength, and foot arch stiffness. The children in the control group will wear traditional footwear with arch support. It is hypothesized that walking with minimalist shoes may impose a positive impact to strengthen the IFM and promote foot arch stiffness for preschool children.

DETAILED DESCRIPTION:
Intrinsic foot muscles(IFM) are the prime stabilizers of the foot. When the IFM become weakened and unstable, the foot and lower limb become more vulnerable to injury. IFM develop across early childhood and evidence suggests that the critical time window for foot arch development is the first 6 years of life (i.e., preschool age). Human's feet and arches developed naturally due to the daily loads imposed on them, while evidence for using protective footwear to promote arch development is very weak. Moreover, the investigation suggested that local children may have a danger in insufficient daily physical activity. Thus the children may be at high risk for having weak feet.

Minimalist shoes are defined as footwear with little to no cushioning, highly flexible soles, and no arch support devices. Minimalist shoes are shaped with a wide toe box, allowing the foot to move more naturally than when confined in conventional footwear. Both running and walking studies have shown that the use of minimalist shoes increases IFM strength by increasing the mechanical load to the foot. Measuring the strength of individual IFM is challenging at best. However, muscle strength has been directly correlated with muscle size. As a result, studies have used imaging techniques such as MRI and ultrasound to measure foot muscle size. A very recent study suggests that walking with minimalist shoes increased the cross-sectional area (CSA), thickness and strength of IFM in adults. Similar findings have been reported by another study adopting a 12-week program.

This study aims to investigate the effects of a 12-week in-school walking training with minimalist shoes for local preschool children on intrinsic foot muscle size, muscle strength, and foot arch stiffness.

In view of the treatment effectiveness and user-friendliness, walking with minimalist shoes may impose a positive impact to strengthen the IFM and promote foot arch stiffness for preschool children.

ELIGIBILITY:
Inclusion Criteria:

* no history of known neurological or orthopedic conditions
* presentation of flexible flatfeet with the Chippaux-Smirak Index >0.6

Exclusion Criteria:

* having previous experience using minimalist footwear
* presenting with any symptoms in the lower limbs within the last three months

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 116 (Estimated)
Dates: Start 2020-12-01 (Estimated); Primary Completion 2022-05-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Cross-sectional area of abductor hallucis in cm^2 | The assessment will be performed at baseline
  An ultrasound scanning unit coupled with a linear array probe will be used to image the cross sectional area of abductor hallucis of the dominant foot.
Cross-sectional area of abductor hallucis in cm^2 | The assessment will be performed at 6 weeks
  An ultrasound scanning unit coupled with a linear array probe will be used to image the cross sectional area of abductor hallucis of the dominant foot.
Cross-sectional area of abductor hallucis in cm^2 | The assessment will be performed at 12 weeks
  An ultrasound scanning unit coupled with a linear array probe will be used to image the cross sectional area of flexor digitorum brevis of the dominant foot.
Cross-sectional area of flexor digitorum brevis in cm^2 | The assessment will be performed at baseline
  An ultrasound scanning unit coupled with a linear array probe will be used to image the cross sectional area of flexor digitorum brevis of the dominant foot.
Cross-sectional area of flexor digitorum brevis in cm^2 | The assessment will be performed at 6 weeks
  An ultrasound scanning unit coupled with a linear array probe will be used to image the cross sectional area of flexor digitorum brevis of the dominant foot.
Cross-sectional area of flexor digitorum brevis in cm^2 | The assessment will be performed at 12 weeks
  An ultrasound scanning unit coupled with a linear array probe will be used to image the cross sectional area of flexor digitorum brevis of the dominant foot.
Thickness of flexor hallucis brevis in cm | The assessment will be performed at baseline
  An ultrasound scanning unit coupled with a linear array probe will be used to image the thickness of flexor hallucis brevis of the dominant foot.
Thickness of flexor hallucis brevis in cm | The assessment will be performed at 6 weeks
  An ultrasound scanning unit coupled with a linear array probe will be used to image the thickness of flexor hallucis brevis of the dominant foot.
Thickness of flexor hallucis brevis in cm | The assessment will be performed at 12 weeks
  An ultrasound scanning unit coupled with a linear array probe will be used to image the thickness of flexor hallucis brevis of the dominant foot.
IFM strength in Newton | The assessment will be performed at baseline
  IFM strength will be measured using a specifically designed dynamometer. Each subject will perform a series of three foot strength tests in a randomized order i.e., doming, hallux flexion, and flexion of the first three lesser toes for the dominant foot. During the data collection, the subjects will be asked to hold the peak force for at least 3 seconds and each test will be performed thrice.
IFM strength in Newton | The assessment will be performed at 6 weeks
  IFM strength will be measured using a specifically designed dynamometer. Each subject will perform a series of three foot strength tests in a randomized order i.e., doming, hallux flexion, and flexion of the first three lesser toes for the dominant foot. During the data collection, the subjects will be asked to hold the peak force for at least 3 seconds and each test will be performed thrice.
IFM strength in Newton | The assessment will be performed at 12 weeks
  IFM strength will be measured using a specifically designed dynamometer. Each subject will perform a series of three foot strength tests in a randomized order i.e., doming, hallux flexion, and flexion of the first three lesser toes for the dominant foot. During the data collection, the subjects will be asked to hold the peak force for at least 3 seconds and each test will be performed thrice.

SECONDARY OUTCOMES:
Foot arch stiffness | The assessment will be performed at baseline, 6 weeks, and 12 weeks
  Walking kinematics and kinetics will be captured for each subject using an eight-camera motion capture system (Vicon, Oxford Metrics Group, Oxford, UK) and a force platform (Kistler Instruments, Winterthur, Switzerland) operating at 200 Hz and 1,000 Hz respectively. Reflective markers will be placed on the first metatarsal head, navicular tuberosity, and medial boarder of the calcaneus of the dominant limb according to a previous study. Following verbal instruction and demonstration, all subjects will be asked to walk barefoot along a 10-meter walkway across the force plate at a self-selected speed. After practicing, five successful walking trials (i.e., within-subject speed < 5% variability) will be obtained from each subject.

CONTACTS AND LOCATIONS:
Overall Officials: Roy TH Cheung, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chen TL, Sze LK, Davis IS, Cheung RT. Effects of training in minimalist shoes on the intrinsic and extrinsic foot muscle volume. Clin Biomech (Bristol). 2016 Jul;36:8-13. doi: 10.1016/j.clinbiomech.2016.05.010. Epub 2016 May 10. PMID 27195735
- [Background] Johnson AW, Myrer JW, Mitchell UH, Hunter I, Ridge ST. The Effects of a Transition to Minimalist Shoe Running on Intrinsic Foot Muscle Size. Int J Sports Med. 2016 Feb;37(2):154-8. doi: 10.1055/s-0035-1559685. Epub 2015 Oct 28. PMID 26509371
- [Background] Ridge ST, Olsen MT, Bruening DA, Jurgensmeier K, Griffin D, Davis IS, Johnson AW. Walking in Minimalist Shoes Is Effective for Strengthening Foot Muscles. Med Sci Sports Exerc. 2019 Jan;51(1):104-113. doi: 10.1249/MSS.0000000000001751. PMID 30113521
- [Background] Ridge ST, Myrer JW, Olsen MT, Jurgensmeier K, Johnson AW. Reliability of doming and toe flexion testing to quantify foot muscle strength. J Foot Ankle Res. 2017 Dec 8;10:55. doi: 10.1186/s13047-017-0237-y. eCollection 2017. PMID 29234467
- [Background] Hollander K, de Villiers JE, Sehner S, Wegscheider K, Braumann KM, Venter R, Zech A. Growing-up (habitually) barefoot influences the development of foot and arch morphology in children and adolescents. Sci Rep. 2017 Aug 14;7(1):8079. doi: 10.1038/s41598-017-07868-4. PMID 28808276